CLINICAL TRIAL: NCT00744627
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Fixed-Dose Study Comparing the Efficacy and Safety of a Single Dose of Lu AA21004 in Acute Treatment of Adults With Generalized Anxiety Disorder
Brief Title: Efficacy and Safety of Vortioxetine (Lu AA21004) for Treatment of Generalized Anxiety Disorder in Adults.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LuAA21004_311; 2008-001766-90 (Registry Identifier: EudraCT); U1111-1112-3487 (Other: WHO)
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-01

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Anxiety Disorders; Drug Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Vortioxetine placebo-matching capsules, orally, once daily for up to 8 weeks.
  Interventions: Drug: Placebo
- Vortioxetine 5 mg (Experimental): Vortioxetine 5 mg, encapsulated tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Encapsulated vortioxetine immediate-release tablets.
  Other Names: Lu AA21004; Brintellix®
  Arms: Vortioxetine 5 mg
Drug: Placebo — Vortioxetine placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of vortioxetine, once daily (QD), in adults with Generalized Anxiety Disorders.

DETAILED DESCRIPTION:
The drug that was tested in this study is called Vortioxetine. Vortioxetine is being tested to treat anxiety in adults who have general anxiety disorder (GAD). This study looked at GAD relief in people who took vortioxetine.

The study enrolled 301 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Vortioxetine 5 mg
* Placebo (dummy inactive pill) - this was a capsule that looked like the study drug but had no active ingredient.

All participants were asked to take one capsule at the same time each day throughout the study.

This multi-center trial was conducted in Europe. The overall time to participate in this study was up to 13 weeks. Participants made 7 visits to the clinic, and were contacted by telephone 4 weeks after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Suffers from a primary diagnosis of Generalized Anxiety Disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria.
* Has a Hamilton Anxiety Scale total score ≥20 at Screening and Baseline.
* Has a Hamilton Anxiety Scale score ≥2 on both Item 1 (anxious mood) and Item 2 (tension) at Screening and Baseline.
* Has a Montgomery-Åsberg Depression Rating Scale total score ≤16 at Screening and Baseline.
* Male and females of childbearing potential who are sexually active agree to use adequate contraception from Screening throughout the duration of the study and for 1 month after the last dose of study medication.

Exclusion Criteria:

* Has received any investigational compound <30 days before Screening or 5 half-lives prior to Screening.
* Has received Lu AA21004 in a previous clinical study or as a therapeutic agent.
* Has 1 or more of the following:

  * Any current psychiatric disorder other than Generalized Anxiety Disorder as defined in the DSM-IV-TR.
  * Current or past history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
  * Any substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR.
  * Presence or history of a clinically significant neurological disorder (including epilepsy).
  * Neurodegenerative disorder (Alzheimer's disease, Parkinson's disease, multiple sclerosis, Huntington disease, etc).
  * Any Axis II disorder that might compromise the study.
* Is required to take excluded medications or it is anticipated that the participant will require treatment with at least 1 of the disallowed concomitant medications during the study including:

  * Nonsteroidal anti-inflammatory drugs
  * Rifampin
  * Macrolide antibiotics
  * Hormones
  * Hypoglycemic agents and Insulin
  * Systemic steroids
  * Antineoplastics
  * Antiobesity agents
  * Antidiarrheal agents (episodic use allowed)
  * Antifungal agents (episodic topical use allowed)
  * Antihistamines (episodic use of loratadine, desloratadine, cetirizine allowed)
  * Cough/cold agents (episodic use allowed but preparations containing pseudoephedrine and narcotics are NOT allowed)
  * Diuretics (episodic use allowed)
* Has a significant risk of suicide according to the investigator's opinion or has a score ≥5 on item 10 (suicidal thoughts) of the Montgomery-Åsberg Depression Rating Scale or has made a suicide attempt in the previous 6 months.
* Has previously failed to respond to adequate treatment with selective serotonin reuptake inhibitors and/or serotonin-norepinephrine reuptake inhibitors.
* Has received electroconvulsive therapy within 6 months prior to Screening.
* Is currently receiving formal cognitive or behavioral therapy, systematic psychotherapy, or plans to initiate such therapy during the study.
* Has a clinically significant unstable illness, for example, hepatic impairment or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, infectious, skin and subcutaneous tissue disorders, or metabolic disturbance.
* Has an alanine aminotransferase, aspartate aminotransferase or bilirubin level >1.5 times the upper limits of normal.
* Has a serum creatinine of >1.5 times the upper limits of normal.
* Has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of study medication. This criterion does not include those participants with basal cell or stage I squamous cell carcinoma of the skin.
* Has clinically significant abnormal vital signs as determined by the investigator.
* Has 1 or more laboratory values outside the normal range, based on the blood or urine samples taken at Screening, that are considered by the investigator to be clinically significant.
* Has thyroid stimulating hormone value outside the normal range at Screening and is deemed clinically significant by the investigator.
* Has an abnormal electrocardiogram as determined by the central reader and confirmed as clinically significant by the investigator.
* Has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy.
* Has previously participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (38):
- Estonia (2):
  - Tallinn
  - Viljandi
- Germany (7):
  - Bad Saarow
  - Berlin
  - Bochum
  - Hüttenberg
  - Rodgau
  - Schwerin
  - Wiesbaden
- Latvia (3):
  - Liepāja
  - Riga
  - Sigulda
- Lithuania (3):
  - Kaunas
  - Palanga
  - Vilnius
- Poland (7):
  - Bialystok
  - Gdynia
  - Gorlice
  - Leszno
  - Skórzewo
  - Torun
  - Tuszyn
- Romania (2):
  - Bucharest
  - Oradea
- Russia (9):
  - Kazan'
  - Lipetsk
  - Moscow
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol
  - Yekaterinburg
- Ukraine (5):
  - Dnipro
  - Kharkiv
  - Liev
  - Luhansk
  - Simferopol

REFERENCES:
- [Result] Bidzan L, Mahableshwarkar AR, Jacobsen P, Yan M, Sheehan DV. Vortioxetine (Lu AA21004) in generalized anxiety disorder: results of an 8-week, multinational, randomized, double-blind, placebo-controlled clinical trial. Eur Neuropsychopharmacol. 2012 Dec;22(12):847-57. doi: 10.1016/j.euroneuro.2012.07.012. Epub 2012 Aug 14. PMID 22898365
- [Derived] Christensen MC, Loft H, Florea I, McIntyre RS. Efficacy of vortioxetine in working patients with generalized anxiety disorder. CNS Spectr. 2019 Apr;24(2):249-257. doi: 10.1017/S1092852917000761. Epub 2017 Oct 30. PMID 29081307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 47 investigative sites in Europe from 23 September 2008 to 07 July 2009.
Pre-assignment Details: Participants with a diagnosis of generalized anxiety disorder were enrolled equally in one of two treatment groups, once a day placebo or 5 mg vortioxetine.
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 5 mg
Started | 151 | 150
Treated | 150 | 150
Completed | 126 | 128
Not Completed | 25 | 22
Not completed — Adverse Event | 6 | 9
Not completed — Lack of Efficacy | 7 | 3
Not completed — Noncompliance | 0 | 1
Not completed — Protocol Deviations | 0 | 2
Not completed — Voluntary Withdrawal | 9 | 6
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 5 mg | Total
Number analyzed (Participants) | 151 | 150 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.49) | 45.0 (14.07) | 45.1 (13.76)
Age, Customized [Number; unit: participants]
  ≤55 years | 112 | 111 | 223
  >55 years | 39 | 39 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 103 | 196
  Male | 58 | 47 | 105
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (White, including Hispanic) | 151 | 150 | 301
  Black | 0 | 0 | 0
  Asian | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian/ Other Pacific Islander | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 8 | 5 | 13
  Non-Hispanic/Non-Latino | 143 | 145 | 288
Region of Enrollment [Number; unit: participants]
  Estonia | 7 | 3 | 10
  Germany | 34 | 37 | 71
  Latvia | 7 | 5 | 12
  Lithuania | 8 | 11 | 19
  Poland | 28 | 31 | 59
  Romania | 5 | 3 | 8
  Russia | 48 | 49 | 97
  Ukraine | 14 | 11 | 25
Weight [Mean (Standard Deviation); unit: kg] | 75.76 (16.370) | 72.97 (14.981) | 74.37 (15.729)
Height [Mean (Standard Deviation); unit: cm] | 169.56 (9.457) | 168.21 (8.653) | 168.89 (9.075)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.29 (4.980) | 25.69 (4.419) | 25.99 (4.710)
Smoking Classification [Number; unit: participants]
  Never Smoked | 99 | 90 | 189
  Current Smoker | 29 | 38 | 67
  Ex-smoker | 23 | 22 | 45
Alcohol Consumption [Number; unit: participants]
  Never | 49 | 47 | 96
  Once monthly or less often | 77 | 72 | 149
  Once a week | 15 | 18 | 33
  2 to 6 times per week | 6 | 10 | 16
  Daily | 4 | 3 | 7
Hamilton Anxiety Scale Total Score [Mean (Standard Deviation); unit: scores on a a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (absent) to 56 (maximum severity).
  scores on a a scale | 26.8 (3.95) | 26.3 (3.92) | 26.6 (3.94)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  scores on a scale | 4.5 (0.67) | 4.5 (0.70) | 4.5 (0.69)
Hospital Anxiety and Depression - Anxiety subscale [Mean (Standard Deviation); unit: scores on a scale] — Hospital Anxiety and Depression (HAD) Anxiety sub-scale consists of 7 items that are assessed on a scale from 0 (no anxiety) to 3 (severe feeling of anxiety). The anxiety subscale determines a state of generalized anxiety including anxious mood, restlessness, anxious thoughts and panic attacks. Scores are summed and range from 0 to 21 (maximal severity).
  scores on a scale | 14.4 (3.08) | 13.8 (2.99) | 14.1 (3.04)
Hospital Anxiety and Depression - Depression subscale [Mean (Standard Deviation); unit: scores on a scale] — Hospital Anxiety and Depression (HAD) Depression sub-scale consists of 7 items that are assessed on a scale from 0 (no depression) to 3 (severe feeling of depression). The depression subscale focuses on the state of lost interest and diminished pleasure response. Scores are summed and range from 0 to 21 (maximal severity).
  scores on a scale | 7.5 (4.03) | 7.6 (3.89) | 7.5 (3.96)
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 12.12 (2.375) | 12.25 (2.219) | 12.18 (2.296)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score at Week 8
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56 where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. Least Squares (LS) means were from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Week 8
Population: The Full Analysis Set included all patients who were randomized, received at least 1 dose of study drug, and had at least 1 post-baseline value for assessment of primary efficacy. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 126 | 128
scores on a scale | -10.49 (0.697) | -14.30 (0.695)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; P-values were tested at the 5% level of significance (ie, statistical significance if P<0.05). To control for multiplicity, a pre-specified sequential testing procedure was applied to compare 5 mg vortioxetine to placebo; as soon as an endpoint was non-significant at 0.05, the testing procedure stopped for all subsequent endpoints; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — Pre-specified sequential statistical testing procedure indicates that when p-value <0.05, hierarchical testing continues; P-values were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis; LS Mean Difference = -3.81, 95% CI 2-sided [-5.74 to -1.88], Standard Error of Mean 0.981

2. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression (HAD) Anxiety Subscale at Week 8
Description: The Hospital Anxiety and Depression (HAD) Anxiety sub-scale consists of 7 items that are assessed on a scale from 0 (no anxiety) to 3 (severe feeling of anxiety). The anxiety subscale determines a state of generalized anxiety including anxious mood, restlessness, anxious thoughts and panic attacks. Scores are summed and range from 0 to 21 (maximal severity). LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 128 | 129
scores on a scale | -4.20 (0.396) | -6.49 (0.393)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; P-values were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis; LS Mean Difference = -2.30, 95% CI 2-sided [-3.39 to -1.20], Standard Error of Mean 0.555

3. Secondary Outcome: Clinical Global Impression Scale-Global Improvement at Week 8
Description: The Clinical Global Impression-Global Improvement scale assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means were from a MMRM with baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 126 | 128
scores on a scale | 2.66 (0.098) | 2.19 (0.098)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; P-values were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis; LS Mean Difference = -0.46, 95% CI 2-sided [-0.73 to -0.19], Standard Error of Mean 0.138

4. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 8
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 109 | 102
scores on a scale | -6.14 (0.631) | -8.10 (0.656)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.031, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; P-values were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis; LS Mean Difference = -1.96, 95% CI 2-sided [-3.74 to -0.18], Standard Error of Mean 0.901

5. Secondary Outcome: Percentage of Responders in HAM-A Total Score at Week 8
Description: Response was defined as participants with a ≥ 50% decrease from Baseline in the Hamilton Anxiety Scale (HAM-A) total score. The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (symptoms absent) to 56 (maximum severity).
Time Frame: Baseline and Week 8
Population: Full analysis set; Last observation carried forward was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 148 | 149
percentage of participants | 39.9 | 61.7
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Logistic regression with explanatory variables for treatment and Baseline HAM-A score; Odds Ratio (OR) = 2.393, 95% CI 2-sided [1.496 to 3.830]

6. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score at Week 8 in Participants With Baseline HAM-A ≥25
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56 where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Week 8
Population: Full analysis set patients with a HAM-A Baseline score ≥25. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 82 | 82
scores on a scale | -10.44 (0.895) | -15.55 (0.904)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; P-values were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis; LS Mean Difference = -5.10, 95% CI 2-sided [-7.61 to -2.60], Standard Error of Mean 1.267

7. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Social Functioning Subscore at Week 8
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The social functioning subscale assesses limitations in social activities because of physical or emotional problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Week 8
Population: The Full Analysis Set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 128 | 129
scores on a scale | 18.02 (1.991) | 26.80 (1.974)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Results presented are for the number of participants at week 8 only; Test type: Superiority or Other; p = 0.002, Mixed model for repeated measurements — SF-36 social functioning subscore was the last endpoint to be tested in the hierarchical testing sequence; P-values were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis; LS Mean Difference = 8.78, 95% CI 2-sided [3.32 to 14.25], Standard Error of Mean 2.774

8. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) Total Score at Other Weeks Assessed
Description: as for outcome 6
Time Frame: Baseline to Weeks 1, 2, 4 and 6.
Population: The Full Analysis Set. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 148 | 149
scores on a scale
  Week 1 (n=146, 148) | -2.46 (0.272) | -2.50 (0.270)
  Week 2 (n=147, 144) | -5.05 (0.407) | -6.21 (0.408)
  Week 4 (n=136, 137) | -7.43 (0.539) | -9.62 (0.538)
  Week 6 (n=128, 129) | -9.17 (0.609) | -11.93 (0.608)

9. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression (HAD) Anxiety Subscale at Other Weeks Assessed
Description: as for outcome 2
Time Frame: Baseline to Weeks 1 and 4
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 148 | 149
scores on a scale
  Week 1 (n=146, 148) | -1.42 (0.226) | -1.14 (0.223)
  Week 4 (n=140, 140) | -3.13 (0.298) | -4.07 (0.296)

10. Secondary Outcome: Clinical Global Impression Scale-Global Improvement at Other Weeks Assessed
Description: as for outcome 3
Time Frame: Baseline to Weeks 1, 2, 4 and 6
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 148 | 149
scores on a scale
  Week 1 (n=146, 148) | 3.58 (0.053) | 3.67 (0.053)
  Week 2 (n=147, 144) | 3.31 (0.070) | 3.10 (0.070)
  Week 4 (n=136, 137) | 2.99 (0.080) | 2.66 (0.080)
  Week 6 (n=128, 129) | 2.74 (0.086) | 2.43 (0.086)

11. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Other Weeks Assessed
Description: as for outcome 4
Time Frame: Baseline to Weeks 1, 2 and 4
Population: Full analysis set where Baseline data were available. A mixed model for repeated measurements (MMRM) based on observed cases was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 124 | 120
scores on a scale
  Week 1 (n=121, 117) | -1.32 (0.314) | -1.12 (0.329)
  Week 2 (n=122, 114) | -2.93 (0.440) | -3.04 (0.459)
  Week 4 (n=112, 107) | -4.35 (0.546) | -5.13 (0.566)

12. Secondary Outcome: Percentage of Responders in HAM-A Total Score at Other Weeks Assessed
Description: as for outcome 5
Time Frame: Baseline and Weeks 1, 2, 4 and 6
Population: Full analysis set; Last observation carried forward was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 148 | 149
percentage of participants
  Week 1 (n=146, 148) | 2.7 | 2.0
  Week 2 (n=148, 149) | 12.2 | 12.1
  Week 4 (n=148, 149) | 20.3 | 28.9
  Week 6 (n=148, 149) | 29.7 | 43.6

13. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score at Other Weeks Assessed in Participants With Baseline HAM-A ≥25
Description: as for outcome 6
Time Frame: Baseline to Weeks 1, 2, 4 and 6
Population: Full analysis set patients with a HAM-A Baseline score ≥25. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 100 | 96
scores on a scale
  Week 1 (n=100, 95) | -2.64 (0.332) | -2.62 (0.341)
  Week 2 (n=99, 92) | -4.89 (0.507) | -6.43 (0.522)
  Week 4 (n=89, 89) | -7.33 (0.694) | -10.08 (0.702)
  Week 6 (n=83, 83) | -9.02 (0.763) | -12.90 (0.771)

14. Secondary Outcome: Percentage of Participants in HAM-A Remission at Each Week Assessed
Description: Remission is defined as a Hamilton Anxiety Scale (HAM-A) total score ≤ 7. The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (symptoms absent) to 56 (maximum severity).
Time Frame: Weeks 1, 2, 4, 6 and 8
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 148 | 149
percentage of participants
  Week 1 (n=146, 148) | 0 | 0
  Week 2 (n=148, 149) | 2.7 | 2.7
  Week 4 (n=148, 149) | 6.8 | 8.7
  Week 6 (n=148, 149) | 12.2 | 16.8
  Week 8 (n=148, 149) | 17.6 | 30.2

15. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Severity of Illness at Each Week Assessed
Description: The Clinical Global Impression-Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Weeks 1, 2, 4, 6 and 8
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 148 | 149
scores on a scale
  Week 1 (n=146, 148) | -0.23 (0.039) | -0.19 (0.039)
  Week 2 (n=147, 144) | -0.53 (0.060) | -0.60 (0.060)
  Week 4 (n=136, 137) | -0.87 (0.071) | -1.04 (0.071)
  Week 6 (n=128, 129) | -1.09 (0.080) | -1.40 (0.080)
  Week 8 (n=126, 128) | -1.26 (0.096) | -1.78 (0.095)

16. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression (HAD) Depression Subscale at Each Week Assessed
Description: The HAD-Depression subscale is completed by the participant and measures depression, focusing on the state of lost interest and diminished pleasure response. The subscale is made up of 7 items that are assessed on a scale from 0 (no depression) to 3 (severe feeling of depression). Participants are required to indicate the response which most accurately reflects the way they have felt over the last few days. The item scores are summed and the total subscore ranges from 0 to 21 (maximal severity). LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Weeks 1, 4 and 8
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 148 | 149
scores on a scale
  Week 1 (n=146, 148) | -0.18 (0.178) | -0.28 (0.176)
  Week 4 (n=140, 140) | -1.08 (0.245) | -1.62 (0.245)
  Week 8 (n=128, 129) | -1.50 (0.297) | -3.18 (0.295)

17. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Social Functioning Subscore at Other Weeks Assessed
Description: as for outcome 7
Time Frame: Baseline to Weeks 2 and 4
Population: The Full Analysis Set with available data at Baseline. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 147 | 149
scores on a scale
  Week 2 (n=147, 149) | 8.50 (1.536) | 8.83 (1.519)
  Week 4 (n=136, 137) | 11.41 (1.773) | 18.45 (1.758)

18. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Physical Functioning Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The physical functioning subscale assesses limitations in physical activities because of health problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 147 | 149
scores on a scale
  Week 2 (n=147, 149) | 2.54 (1.160) | 3.39 (1.146)
  Week 4 (n=136, 137) | 2.15 (1.149) | 8.34 (1.137)
  Week 8 (n=128, 129) | 4.48 (1.271) | 10.69 (1.258)

19. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Role-Physical Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The role-physical subscale assesses limitations in usual role activities because of physical health problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 147 | 149
scores on a scale
  Week 2 (n=147, 149) | 4.72 (1.488) | 5.99 (1.474)
  Week 4 (n=136, 137) | 6.89 (1.592) | 11.89 (1.578)
  Week 8 (n=128, 129) | 8.96 (1.897) | 18.39 (1.880)

20. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Bodily Pain Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The bodily pain sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 147 | 149
scores on a scale
  Week 2 (n=147, 149) | 6.49 (1.702) | 7.40 (1.681)
  Week 4 (n=136, 137) | 6.81 (1.875) | 10.62 (1.856)
  Week 8 (n=128, 129) | 10.90 (1.903) | 15.38 (1.883)

21. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) General Health Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The general health sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 147 | 149
scores on a scale
  Week 2 (n=147, 149) | 4.54 (0.992) | 6.04 (0.979)
  Week 4 (n=136, 137) | 8.45 (1.292) | 10.36 (1.280)
  Week 8 (n=128, 129) | 9.76 (1.409) | 16.30 (1.396)

22. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Vitality Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The vitality sub-score assesses energy and fatigue, and ranges from 0 (best) - 100 (worst). LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 147 | 149
scores on a scale
  Week 2 (n=147, 149) | 5.44 (1.275) | 8.11 (1.261)
  Week 4 (n=136, 137) | 8.36 (1.500) | 13.38 (1.486)
  Week 8 (n= 128, 129) | 12.56 (1.686) | 22.53 (1.671)

23. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Role-Emotional Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The role-emotional subscale assesses limitations in usual role activities because of emotional problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 147 | 149
scores on a scale
  Week 2 (n=147, 149) | 7.27 (1.480) | 9.62 (1.463)
  Week 4 (n=136, 137) | 13.41 (1.871) | 19.04 (1.856)
  Week 8 (n=128, 129) | 18.96 (2.138) | 28.13 (2.121)

24. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Mental Health Subscore at Each Week Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The mental health sub-score assesses general mental health (psychological distress and well-being) and ranges from 0 (best) - 100 (worst). LS means were from a MMRM with Baseline-by-week, center, week and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Weeks 2, 4 and 8
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 147 | 149
scores on a scale
  Week 2 (n=147, 149) | 5.58 (1.166) | 8.90 (1.152)
  Week 4 (n=136, 137) | 9.79 (1.432) | 14.73 (1.421)
  Week 8 (n=128, 129) | 13.51 (1.693) | 21.75 (1.681)

25. Secondary Outcome: Health Care Resource Utilization as Assessed by the Health Economic Assessment Questionnaire
Description: Healthcare resource utilization was assessed by the Health Economic Assessment (HEA) questionnaire, which monitors the participants absenteeism from work, as well as resource use such as visits to a general practitioner, outpatient and inpatient services, hospitalization, medications, and other relevant services over the past 8 weeks.
Time Frame: Baseline and Week 8
Population: Full analysis set.
Measure: Number; unit: participants
Arm/Group | Placebo | Vortioxetine 5 mg
Number analyzed (Participants) | 148 | 149
participants
  Baseline: Any resource use | 79 | 84
  Baseline: Any hospitalization-related services | 7 | 3
  Baseline: Hospitalization related to anxiety | 4 | 2
  Baseline: Any sick leave | 7 | 7
  Baseline: Sick leave related to anxiety | 4 | 4
  Week 8: Any resource use | 14 | 25
  Week 8: Any hospitalization-related service | 0 | 1
  Week 8: Hospitalization related to anxiety | 0 | 0
  Week 8: Any sick leave | 2 | 4
  Week 8: Sick leave related to anxiety | 2 | 3

ADVERSE EVENTS:
Time Frame: Safety was assessed during the 8-week treatment period and a 4-week follow-up period.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vortioxetine 5 mg
Serious Adverse Events (participants affected / at risk) | 1/150 | 0/150
Other Adverse Events (participants affected / at risk) | 36/150 | 48/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=150) | Vortioxetine 5 mg (N=150)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=150) | Vortioxetine 5 mg (N=150)
Nausea (Gastrointestinal disorders) | 9 | 18
Dry mouth (Gastrointestinal disorders) | 4 | 5
Vomiting (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Fatigue (General disorders) | 4 | 1
Nasopharyngitis (Infections and infestations) | 1 | 5
Bronchitis (Infections and infestations) | 4 | 0
Influenza (Infections and infestations) | 1 | 3
Headache (Nervous system disorders) | 13 | 12
Dizziness (Nervous system disorders) | 4 | 9
Somnolence (Nervous system disorders) | 2 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.